CLINICAL TRIAL: NCT06843655
Title: Radiological Markers in Locally Advanced Rectal Cancer
Acronym: LARC
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Francesco De Cobelli, Principal Investigator, MD, IRCCS San Raffaele
Other Study IDs: LARC Protocol
Record Dates: First submitted 2025-02-18; First posted 2025-02-25 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Locally Advanced Rectal Carcinoma
Keywords: Locally Advanced Rectal Cancer (LARC); Total Neoadjuvant Therapy (TNT); Diffusion-Weighted MRI (DWI); Likert Score; Radiological Prognostic Markers

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this observational study is to evaluate the prognostic significance of radiological markers, including the Likert Score derived from diffusion-weighted MRI (DWI), in patients with locally advanced rectal cancer (LARC) treated with total neoadjuvant therapy (TNT). Specifically, the study investigates the association between the Likert Score on restaging MRI and key clinical outcomes, such as overall survival (OS) and time to progression (TTP). Furthermore, it examines the impact of other MRI-derived markers-extramural venous invasion (EMVI), tumor deposits (TDs), and mesorectal fascia invasion (MFI)-on disease progression and patient prognosis. This study retrospectively analyzes 179 patients who underwent TNT followed by surgery between 2009 and 2022. Participants were required to have pre- and post-treatment MRI scans. MRI imaging data and patient outcomes, including overall survival (OS) and time to progression (TTP), will be analyzed over a follow-up period extending until July 31, 2024. Findings from this study may help refine MRI-based prognostic tools for personalized treatment strategies in rectal cancer.

DETAILED DESCRIPTION:
This study investigates the prognostic role of diffusion-weighted MRI (DWI), using the Likert Score and other radiological markers, in patients with locally advanced rectal cancer (LARC) undergoing total neoadjuvant therapy (TNT) followed by radical surgery. The study cohort consists of 179 patients who received TNT between 2009 and 2022 at our institution. Inclusion criteria required patients to have biopsy-confirmed stage II-III LARC, available MRI at both staging and restaging time points, and completion of the TNT protocol.

The TNT regimen included up to three cycles of modified XELOX chemotherapy (oxaliplatin and capecitabine), with the first cycle administered as induction chemotherapy and the remaining two cycles administered concurrently with radiotherapy (total dose: 46.2 Gy in 18 fractions). Surgical resection was performed at a median of 11 weeks post-radiotherapy, with adjuvant chemotherapy administered based on histopathology findings.

MRI acquisition was standardized using a 1.5-T scanner, with DWI sequences applied to assess key prognostic markers, including extramural venous invasion (EMVI), tumor deposits (TDs), and mesorectal fascia invasion (MFI). The Likert Score, a five-point grading system based on DWI findings, was applied to restaging MRI to stratify treatment response, with scores of 0-2 indicating a favorable response and 3-4 indicating a poor response.

The study's primary objective is to evaluate the impact of the Likert Score on overall survival (OS) and time to progression (TTP). Secondary objectives include assessing the prognostic significance of EMVI, TDs, and MFI in predicting OS and TTP. The statistical analysis will include Kaplan-Meier survival curves to estimate OS and TTP, stratified according to the presence/score of radiological markers, Cox proportional hazards regression to assess the impact of prognostic factors on survival outcomes, Fisher's exact test to evaluate associations between categorical variables, and Cohen's Kappa to measure interobserver agreement in MRI assessments..

This study aims to refine MRI-based prognostic assessment tools to enhance personalized treatment strategies for rectal cancer. Findings from this research may support the integration of DWI-based Likert Score evaluation into clinical practice to improve risk stratification and treatment decision-making in patients with LARC undergoing TNT. The follow-up period extends until July 31, 2024, ensuring a comprehensive analysis of long-term outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Risonanza Magnetica informed consent signed
* All patients that received total neoadjuvant therapy (TNT) (chemo/radiotherapy followed by surgery), between 2009 and 2022 at our institution
* Staging and re-staging MRI available

Exclusion Criteria:

* Staging and re-staging MRI not available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study includes patients with locally advanced rectal cancer (LARC) who underwent total neoadjuvant therapy (TNT) followed by surgery at our institution between 2009 and 2022. MRI imaging was performed both at initial staging and after TNT before surgery. The follow-up period extends until July 31, 2024, with survival outcomes being analyzed retrospectively.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Time To Progression (TTP) Stratified by Likert Score | 5 years
  TTP will be measured as the time from diagnosis to disease progression, as assessed through clinical, radiological, or pathological criteria. Patients will be stratified based on the Likert Score derived from diffusion-weighted MRI (DWI) at restaging. Kaplan-Meier survival curves will be used to estimate progression-free probabilities, with comparisons between groups performed using the log-rank test. Cox proportional hazards regression will be used to evaluate the prognostic significance of the Likert Score. TTP will be measured in months, defined as the time from diagnosis to documented disease progression based on clinical, radiological, or pathological criteria.
Overall Survival (OS) Stratified by Likert Score | 5 years
  OS will be measured as the time from diagnosis to death from any cause in patients with locally advanced rectal cancer (LARC) treated with total neoadjuvant therapy (TNT). Patients will be stratified based on the Likert Score derived from diffusion-weighted MRI (DWI) at restaging. Kaplan-Meier survival curves will be used to estimate survival probabilities, and differences between groups will be compared using the log-rank test. Cox proportional hazards regression will be performed to assess the prognostic value of the Likert Score. OS will be measured in months, defined as the time from diagnosis to death. Patients alive at the end of the study period or lost to follow-up will be censored at their last recorded visit.

SECONDARY OUTCOMES:
Prognostic Value of EMVI Score on Time to Progression (TTP) | 5 years
  The study will evaluate the impact of extramural venous invasion (EMVI) on time to progression (TTP) in patients with locally advanced rectal cancer (LARC) undergoing total neoadjuvant therapy (TNT). TTP, measured in months, will be defined as the time from diagnosis to documented disease progression based on clinical, radiological, or pathological criteria. Patients will be stratified by EMVI Score, assessed on staging MRI. Progression-free probabilities will be estimated using Kaplan-Meier survival curves, with group comparisons performed via the log-rank test. The prognostic value of the EMVI Score will be examined through Cox proportional hazards regression.
Prognostic Value of Tumor Deposits on Time to Progression (TTP) | 5 years
  The study will evaluate the impact of tumor deposits (TDs) on time to progression (TTP) in patients with locally advanced rectal cancer (LARC) undergoing total neoadjuvant therapy (TNT). TTP, measured in months, will be defined as the time from diagnosis to documented disease progression based on clinical, radiological, or pathological criteria. Patients will be stratified based on the presence of TDs, identified on staging MRI. Progression-free probabilities will be estimated using Kaplan-Meier survival curves, with group comparisons performed via the log-rank test. The prognostic significance of TDs will be analyzed using Cox proportional hazards regression.
Prognostic Value of Mesorectal Fascia Infiltration on Time to Progression (TTP) | 5 years
  The study will evaluate the impact of mesorectal fascia infiltration (MFI) on time to progression (TTP) in patients with locally advanced rectal cancer (LARC) undergoing total neoadjuvant therapy (TNT). TTP, measured in months, will be defined as the time from diagnosis to documented disease progression based on clinical, radiological, or pathological criteria. Patients will be stratified based on the presence of MFI, identified on staging MRI. Progression-free probabilities will be estimated using Kaplan-Meier survival curves, with group comparisons performed via the log-rank test. The prognostic significance of MFI will be analyzed using Cox proportional hazards regression.
Prognostic Value of EMVI Score on Overall Survival (OS) | 5 years
  The study will evaluate the impact of the EMVI Score on OS in patients with locally advanced rectal cancer (LARC) undergoing total neoadjuvant therapy (TNT). OS, measured in months, will be defined as the time from diagnosis to death. Patients will be stratified by EMVI Score, assessed on staging MRI. Survival probabilities will be estimated using Kaplan-Meier curves, with group comparisons performed via the log-rank test. The prognostic significance of the EMVI Score will be analyzed using Cox proportional hazards regression.
Prognostic Value of Tumor Deposits on Overall Survival (OS) | 5 years
  The study will evaluate the impact of tumor deposits (TDs) on OS in patients with locally advanced rectal cancer (LARC) undergoing total neoadjuvant therapy (TNT). OS, measured in months, will be defined as the time from diagnosis to death. Patients will be stratified based on the presence of TDs, identified on staging MRI. Survival probabilities will be estimated using Kaplan-Meier curves, with group comparisons performed via the log-rank test. The prognostic significance of TDs will be analyzed using Cox proportional hazards regression.
Prognostic Value of Mesorectal Fascia Infiltration on Overall Survival (OS) | 5 years
  The study will evaluate the impact of mesorectal fascia infiltration (MFI) on OS in patients with locally advanced rectal cancer (LARC) undergoing total neoadjuvant therapy (TNT). OS, measured in months, will be defined as the time from diagnosis to death. Patients will be stratified based on the presence of MFI, assesed on staging MRI. Survival probabilities will be estimated using Kaplan-Meier curves, with group comparisons performed via the log-rank test. The prognostic significance of MFI will be analyzed using Cox proportional hazards regression.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Radiology, IRCCS Ospedale San Raffaele, Milan, Italy

IPD SHARING:
Plan to Share IPD: No